CLINICAL TRIAL: NCT02638571
Title: Evaluation of the Effectiveness of Nutrition Education Intervention Among Rural Mothers on Pulse and Cereal Mix Complementary Food and Nutritional Status of Children Age 6-24 Months in Sidama Zone, Southern Ethiopia
Brief Title: Evaluation Nutrition Education Intervention on Pulse and Cereal Mix for Complementary Food in Southern Ethiopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Hawassa University (Other)
Responsible Party: Principal Investigator, Carol J. Henry, Ph.D., University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PULSE-HEW
Record Dates: First submitted 2015-12-18; First posted 2015-12-23 (Estimated); Last update posted 2024-05-08 (Actual); Status verified 2018-10

CONDITIONS: Dietary Habits; Health Knowledge, Attitudes, Practices; Wasting
MeSH Terms: conditions — Feeding Behavior; Behavior; Cachexia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual education (Sham Comparator): Households in the control clusters (kebeles) will receive usual nutrition education from Health extension workers, about complementary foods, over 9 months.
  Interventions: Other: enhanced education on pulse use in complementary foods
- Enhanced Education (Experimental): Additional education sessions from Health extension workers (HEWs) trained on use of pulses for complementary foods (CF). HEWs provide nutrition education programs and counseling about pulse-cereal mix complementary foods, over 9 months.
  Interventions: Other: enhanced education on pulse use in complementary foods

INTERVENTIONS:
Other: enhanced education on pulse use in complementary foods — Enhanced Nutrition education with sessions and counseling by health extension workers

SUMMARY:
The overall purpose of the study is to evaluate nutrition education interventions to promote pulse incorporated complementary food to the wider rural community through the government system to improve maternal knowledge, attitude and practice (KAP) and nutritional status of young children (6 to 24 months). The hypothesis is that nutrition education improves mothers knowledge, attitude and practice of pulse incorporated complementary food and improves dietary intake of iron and zinc and nutritional status of young children.

DETAILED DESCRIPTION:
Only 9% of the population in Southern Ethiopia consumes pulse and pulse total contribution of the diet is less than 4.9% for women and less than 3.3% for children.Young children are at risk of developing malnutrition because of dietary inadequacy. Educational interventions can improve feeding practices and growth of young children. The overall purpose of the study is to evaluate nutrition education interventions to promote pulse incorporated complementary food to the wider rural community through the government system to improve maternal knowledge, attitude and practice (KAP) and nutritional status of young children (6 to 24 months). The hypothesis is that nutrition education improves mothers knowledge, attitude and practice of pulse incorporated complementary food and improves dietary intake of iron and zinc and nutritional status of young children. Before, at midline and end of the intervention we will assess the KAP of mothers, dietary intake of iron and zinc and nutritional status of young children. The nutrition education intervention will be given for 9 months. Serum ferritin, serum zinc, C-Reactive protein and hemoglobin and dietary intake of iron and zinc of young children will be measured at the beginning and ending of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-15 months
* Apparently healthy
* Being breastfed at time of recruitment
* The mothers are permanent residents of the kebele

Exclusion Criteria:

* Infant undergoing treatment with supplemental foods for malnutrition

Ages: 6 Months to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 772 (Actual)
Dates: Start 2016-01-19 (Actual); Primary Completion 2016-11-22 (Actual); Study Completion 2016-11-22 (Actual)

PRIMARY OUTCOMES:
Maternal knowledge, attitudes and practices towards pulse-cereal mix complementary food | 9 months
  Using validated questions on knowledge, attitude and practices

SECONDARY OUTCOMES:
Weight for height Z-score of children | 9 months
  Change in z-score of measured weight and measured height (length) ratio at 9 months
Zinc status of children | 9 months
  Measurement of serum zinc against WHO standards
Iron status | 9 months
  iron status as determined by serum ferritin corrected for inflammation using markers, whole hemoglobin to define anemia status using WHO standards.

CONTACTS AND LOCATIONS:
Overall Officials: Carol J Henry, PhD, Principal Investigator — University of Saskatchewan

IPD SHARING:
Plan to Share IPD: No
Only mean (or median) data will be published. If there are correlations or regressions the r or r2 will be published

REFERENCES:
- [Background] Amare B, Moges B, Fantahun B, Tafess K, Woldeyohannes D, Yismaw G, Ayane T, Yabutani T, Mulu A, Ota F, Kassu A. Micronutrient levels and nutritional status of school children living in Northwest Ethiopia. Nutr J. 2012 Dec 13;11:108. doi: 10.1186/1475-2891-11-108. PMID 23237638
- [Background] Bhutta ZA, Das JK, Rizvi A, Gaffey MF, Walker N, Horton S, Webb P, Lartey A, Black RE; Lancet Nutrition Interventions Review Group, the Maternal and Child Nutrition Study Group. Evidence-based interventions for improvement of maternal and child nutrition: what can be done and at what cost? Lancet. 2013 Aug 3;382(9890):452-477. doi: 10.1016/S0140-6736(13)60996-4. Epub 2013 Jun 6. PMID 23746776
- [Background] Hirvone K, & Hoddinot J. Agricultural production and children's diets: Evidence from rural Ethiopia. EDRI & IFPRI, working paper 69.
- [Background] Kebebu A, Whiting S, & Henry C. Formulation of a complementary food fortified with broad beans (vicia faba) in Southern Ethiopia. African Journal of Food, Agriculture, Nutrition and Development. 2013; 13(3): 7789-7803.
- [Background] Kuma T. Analysis of changes in Food Consumption Pattern in Urban Ethiopia. EDRI. 2010.
- [Background] Negash C, Belachew T, Henry CJ, Kebebu A, Abegaz K, Whiting SJ. Nutrition education and introduction of broad bean-based complementary food improves knowledge and dietary practices of caregivers and nutritional status of their young children in Hula, Ethiopia. Food Nutr Bull. 2014 Dec;35(4):480-6. doi: 10.1177/156482651403500409. PMID 25639132
- [Background] Tefera T. Determinants of smallholder pulse producers market orientation in Southern Ethiopia. Asian Journal of Business Management. 2014; 6(2); 97-103.
- [Result] Berhanu G, Henry CJ, Whiting SJ, Green TJ. 2017 Assessment of knowledge, attitude and practice of mothers on pulse incorporated complementary food and its correlations with diet diversity and nutritional status of their children aged 6-15 months in two rural districts of Sidama, South Ethiopia. International Journal of Nutritional Sciences (Special Issue on Malnutrition). 2(1): id1017 (2017).
- [Derived] Teshome GB, Whiting SJ, Green TJ, Mulualem D, Henry CJ. Scaled-up nutrition education on pulse-cereal complementary food practice in Ethiopia: a cluster-randomized trial. BMC Public Health. 2020 Sep 22;20(1):1437. doi: 10.1186/s12889-020-09262-8. PMID 32962685